CLINICAL TRIAL: NCT00770159
Title: A Double-Blind, Placebo-Controlled, Once-Weekly, Multiple-Dose Study to Investigate the Safety, Tolerability, Plasma Concentration Profile and Effects on Biochemical Markers of Bone Resorption of MK0822 in Healthy Postmenopausal Female Subjects
Brief Title: A Study to Test Once-Weekly Doses of Odanacatib (MK0822) on Healthy Adult Females (0822-005)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-005; MK0822-005; 2008_559
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MK0822
  Interventions: Drug: odanacatib
- 2 (Placebo Comparator): Placebo to MK0822
  Interventions: Drug: Comparator: placebo to MK0822

INTERVENTIONS:
Drug: odanacatib — Panel A: MK0822 tablets 25 mg once weekly for 3 weeks. Panel B: MK0822 tablets 50 mg once weekly for 3 weeks. Panel C: MK0822 tablets 100 mg once weekly for 3 weeks. Panel D: MK0822 tablets 5 mg once weekly for 3 weeks. Panel E: MK0822 tablets 100 mg once weekly for 6 weeks.
  Arms: 1
Drug: Comparator: placebo to MK0822 — Panel A: placebo to MK0822 tablets 25 mg once weekly for 3 weeks. Panel B: placebo to MK0822 tablets 50 mg once weekly for 3 weeks. Panel C: placebo to MK0822 tablets 100 mg once weekly for 3 weeks. Panel D: placebo to MK0822 tablets 5 mg once weekly for 3 weeks. Panel E: placebo to MK0822 tablets 100 mg once weekly for 6 weeks.
  Arms: 2

SUMMARY:
This study will assess the safety, tolerability, PK, and PD of a once weekly dose of MK0822 in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Subject is less than or equal to 75 years of age
* Subject is a postmenopausal female
* Subject is within 30% of ideal body weight
* Subject is judged to be in good health
* Subject is a nonsmoker
* Subject is willing to avoid excessive alcohol consumption for the duration of the study
* Subject is willing to avoid strenuous physical activity for the duration of the study
* Subject agrees to refrain from consuming grapefruit or grapefruit juice for the duration of the study

Exclusion Criteria:

* Subject has a history of multiple/severe allergies to foods or drugs
* Subject has had surgery within 12 weeks of starting study or has given blood within 4 weeks of starting study
* Subject has a history of major GI abnormalities/ulcers, or genitourinary, cardiovascular, hepatic, pulmonary, psychiatric, endocrine, or metabolic diseases
* Subject has a history of bone disease or treatment with bisphosphonates
* Subject has an infection/condition that would suppress the immune system, including HIV
* Subject has a history of chronic/active hepatic (liver) disease, including Hepatitis B and C
* Subject regularly uses illegal drugs
* Subject consumes more than 3 alcoholic beverages per day
* Subject consumes more than 4 cups of brewed coffee (or equivalent caffeinated beverages) per day
* Subject requires use of any prescription or non-prescription medications during the study
* Part I only: subject has received treatment with any of the following: any estrogen preparation, anabolic steroids, calcitonin, or progestins within 6 months of study start; thyroid hormone if not on a stable dose; fluoride treatment greater than 1mg/day for more than 2 weeks; Glucocorticoid treatment; Vitamin A greater than 10,000 U/day, vitamin D greater than 2000 U/day, anticonvulsants; selective estrogen receptor modulators within 6 months of study start; parathyroid hormone within 2 years of study start; or bisphosphonates.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With One or More Adverse Events | Up to 7 weeks
Number of Participants Who Discontinued Study Drug Due to Adverse Events | Up to 6 weeks

SECONDARY OUTCOMES:
Area Under Time Curve From 0 to 24 Hours (AUC 0-24hr) at Week 1 and Week 3 | Up to 24 hours postdose, Week 1 and Week 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Stoch SA, Zajic S, Stone J, Miller DL, Van Dyck K, Gutierrez MJ, De Decker M, Liu L, Liu Q, Scott BB, Panebianco D, Jin B, Duong LT, Gottesdiener K, Wagner JA. Effect of the cathepsin K inhibitor odanacatib on bone resorption biomarkers in healthy postmenopausal women: two double-blind, randomized, placebo-controlled phase I studies. Clin Pharmacol Ther. 2009 Aug;86(2):175-82. doi: 10.1038/clpt.2009.60. Epub 2009 May 6. PMID 19421185